CLINICAL TRIAL: NCT03231423
Title: Effect of Drain Usage on Patient Comfort on Laparoscopic Gastric Bypass Surgery
Brief Title: Effect of Drainage on Laparoscopic Gastric Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ersin Gündoğan, Operator doctor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/181
Record Dates: First submitted 2017-07-12; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Obesity, Morbid
Keywords: Obesity; VAS; Pain; Laparoscopy; Bypass
MeSH Terms: conditions — Obesity, Morbid; Obesity; Pain | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DRAIN PLACEMENT (Experimental): Effects of drainage
  Interventions: Other: Drainage
- DRAIN NOT PLACED (No Intervention): Effects of not using drain

INTERVENTIONS:
Other: Drainage — Using drain after operation
  Arms: DRAIN PLACEMENT

SUMMARY:
Introduction RYGB surgeon; Have become increasingly morbid obesity treatment methods with improvements in minimally invasive surgery. Ensuring patient comfort and early return to life are the criteria that should be given priority in this treatment method. The purpose of this study is to determine the use of drain, which closely affects these criteria; And the effect on patient comfort.

DETAILED DESCRIPTION:
Question the necessity of routine use of drain in RYGB surgeon

ELIGIBILITY:
Inclusion Criteria:

* Morbid obese patients

Exclusion Criteria:

* Cirrhotic patients, those under 18 years of age, additional intraabdominal surgeries during LRYGBP and those who had previously undergone obesity surgery (revision surgery) were excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
3-Item Pain Intensity measyre (P3) | 8 months
  self reported pain intensity morning, second day and third day. Each item is scored 0-10 ( 0: no pain- 10: pain as bad as can be)

IPD SHARING:
Plan to Share IPD: No